CLINICAL TRIAL: NCT05144737
Title: A Virtual Cardiometabolic Health Program for African Immigrants: The Afro-DPP Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: IRB00251726; 129674 (Other Grant/Funding Number: National Institute For Nursing Research)
Record Dates: First submitted 2021-11-22; First posted 2021-12-03 (Actual); Last update posted 2024-08-23 (Actual); Status verified 2024-08

CONDITIONS: Diabetes Mellitus; Diabetes Mellitus, Type 2; PreDiabetes; Hypertension; High Blood Pressure; High Blood Sugar; Obesity; Overweight; Overweight and Obesity; Overweight or Obesity
Keywords: African immigrant; Prediabetes; National Diabetes Prevention Program
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2; Prediabetic State; Hypertension; Hyperglycemia; Obesity; Overweight

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immediate Intervention Group (Other): Participants in the immediate intervention group will immediately begin 6 months of the adapted DPP lifestyle intervention with a Lifestyle Coach and remote monitoring of blood pressure and body composition. This will be followed by a 6-month observation period where the intervention (Lifestyle Coach) will be withdrawn. In this period, participants will be evaluated for the maintenance of lifestyle changes.
  Interventions: Behavioral: The Diabetes Prevention Program
- Delayed Intervention Group (Other): Participants in the delayed intervention group will receive remote monitoring of blood pressure and body composition for the 1st 6 months (without the Lifestyle Coach) and then will receive the adapted DPP lifestyle intervention with a Lifestyle Coach after 6 months.
  Interventions: Behavioral: The Diabetes Prevention Program

INTERVENTIONS:
Behavioral: The Diabetes Prevention Program — The multicomponent intervention will focus on intensive lifestyle modification delivered by the Lifestyle Coach. The Lifestyle Coach of African origin will be responsible for delivering the intensive lifestyle intervention and implementing the adapted diabetes prevention program (DPP) curriculum.

SUMMARY:
A pilot study titled "A Virtual Cardiometabolic Health Program for African Immigrants (The Afro-DPP Program) will be conducted to address the cardiometabolic of community-dwelling African immigrants who have multiple cardiometabolic risk factors including hypertension, Type 2 Diabetes, high cholesterol, and overweight/obesity. The proposed study will recruit a total of 60 participants and will use a non-equivalent control group design to test the effectiveness of the intervention at two African churches in the Baltimore, Washington, D.C. area. The two churches will be randomly assigned to the intervention or delayed intervention group. At the end of a 6-month follow-up period, the control church will receive the intervention (delayed control group). All participants will receive a Bluetooth-enabled digital scale (Omron Model: BCM-500) that measures body composition including Body Weight, Body Fat percentage, Visceral Fat, Skeletal Muscle percentage, Resting Metabolism and Body Mass Index. A Bluetooth-enabled blood pressure monitor (Omron Model: BP7250) will also be distributed to all participants. All participants will download the Omron Connect app which will allow the participants to sync participants' blood pressure readings and body composition readings into the app. The research team will access these readings to monitor study outcomes and participants progress during the follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* African immigrants who are aged 25-75 years
* Participants who report being uninsured or have no access to a healthcare provider
* Have at least two of the following chronic conditions:
* Body-mass index ≥ 25 kg/m2
* Self-reported fasting plasma glucose of 95 to 125 mg/d or HbA1c of 5.7-6.5% in the past 6 months
* Systolic blood pressure ≥140 mmHg or diastolic blood pressure ≥ 90 mmHg

Exclusion Criteria:

* Participants who cannot communicate in English
* Participants who have cognitive challenges that would restrict them from participation
* Participants who have any serious illness that would interfere with participation
* Participants who are not members of the churches that are involved in this study

Ages: 25 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-11-21 (Actual); Primary Completion 2024-08-16 (Actual); Study Completion 2024-08-16 (Actual)

PRIMARY OUTCOMES:
Change in systolic blood pressure over a 6-month period | Baseline, 1 month, 3 months, 6 months
  A Bluetooth-enabled blood pressure monitor (Omron Model: BP7250) will be distributed to all participants. All participants will download the Omron Connect app which will allow them to sync their systolic blood pressure readings (mmHg) into the app.
Change in diastolic blood pressure over a 6-month period | Baseline, 1 month, 3 months, 6 months
  A Bluetooth-enabled blood pressure monitor (Omron Model: BP7250) will be distributed to all participants. All participants will download the Omron Connect app which will allow them to sync their diastolic blood pressure readings (mmHg) into the app.
Change in body weight over a 6-month period | Baseline, 1 month, 3 months, 6 months
  All participants will receive a Bluetooth-enabled digital scale (Omron Model: BCM-500) that measures body weight (Kg).
Change in body fat percentage over a 6-month period | Baseline, 1 month, 3 months, 6 months
  All participants will receive a Bluetooth-enabled digital scale (Omron Model: BCM-500) that measures body fat percentage (%).
Change in visceral fat over a 6-month period | Baseline, 1 month, 3 months, 6 months
  All participants will receive a Bluetooth-enabled digital scale (Omron Model: BCM-500) that measures Visceral Fat (rating levels 1-59).
Change in skeletal muscle percentage over a 6-month period | Baseline, 1 month, 3 months, 6 months
  All participants will receive a Bluetooth-enabled digital scale (Omron Model: BCM-500) that measures Skeletal Muscle percentage (%).
Change in resting metabolism over a 6-month period | Baseline, 1 month, 3 months, 6 months
  All participants will receive a Bluetooth-enabled digital scale (Omron Model: BCM-500) that measures Resting Metabolism (kcal).
Change in body mass index over a 6-month period | Baseline, 1 month, 3 months, 6 months
  All participants will receive a Bluetooth-enabled digital scale (Omron Model: BCM-500) that measures Body Mass Index (Kg/m^2).

SECONDARY OUTCOMES:
Change in global cardiovascular disease risk | Baseline, 6 months and 12 months
  Global cardiovascular disease (CVD) risk will be calculated using the body mass index-based cardiovascular risk score. Higher scores indicate higher CVD risk. Continuous risk scores will be used to classify patients into risk categories according to the Adult Treatment Panel III of the National Cholesterol Education Program (ATPIII): low (<10%), moderate (10-20%), and high (>20%).
Change in body mass index over a 12-month period | Baseline and 12 months
  Body mass index (Kg/m^2) will be calculated using the adult body mass index calculator provided by Centers for Disease Control and Prevention.
Change in systolic blood pressure over a 12-month period | Baseline and 12 months
  A Bluetooth-enabled blood pressure monitor (Omron Model: BP7250) will be distributed to all participants. All participants will download the Omron Connect app which will allow them to sync their systolic blood pressure readings (mmHg) into the app.
Change in diastolic blood pressure over a 12-month period | Baseline and 12 months
  A Bluetooth-enabled blood pressure monitor (Omron Model: BP7250) will be distributed to all participants. All participants will download the Omron Connect app which will allow them to sync their diastolic blood pressure readings (mmHg) into the app.
Change in body weight over a 12-month period | Baseline and 12 months
  All participants will receive a Bluetooth-enabled digital scale (Omron Model: BCM-500) that measures body weight (Kg).
Change in body fat percentage over a 12-month period | Baseline and 12 months
  All participants will receive a Bluetooth-enabled digital scale (Omron Model: BCM-500) that measures body fat percentage (%).
Change in visceral fat over a 12-month period | Baseline and 12 months
  All participants will receive a Bluetooth-enabled digital scale (Omron Model: BCM-500) that measures Visceral Fat (rating levels 1-59).
Change in skeletal muscle percentage over a 12-month period | Baseline and 12 months
  All participants will receive a Bluetooth-enabled digital scale (Omron Model: BCM-500) that measures Skeletal Muscle percentage (%).
Change in resting metabolism over a 12-month period | Baseline and 12 months
  All participants will receive a Bluetooth-enabled digital scale (Omron Model: BCM-500) that measures Resting Metabolism (kcal).

OTHER OUTCOMES:
Change in quality of life over the 12-month period | Baseline, 6 months and 12 months
  A validated tool by the name of PROMIS global measure will be provided by the Patient-Reported Outcomes Measurement Information System (PROMIS). This 9 items on this tool will measure the participants' fatigue, emotional distress, social health, and physical function. The 9 of the 10 PROMIS global measure items will be scored on a Likert scale from 1 to 5, with 5 representing the best health. Higher scores from summation of the nine items indicate better quality of life.
Change in pain severity over the 12-month period | Baseline, 6 months and 12 months
  A validated tool by the name of PROMIS global measure will be provided by the Patient-Reported Outcomes Measurement Information System. One item on this tool will measure the participants' perception of pain. The pain item uses a response scale of 0-10, which will be rescored to a 5-point scale. Higher scores on the Pain item indicate higher pain severity.

CONTACTS AND LOCATIONS:
Overall Officials: Yvonne Commodore-Mensah, PhD, MSH, RN, Principal Investigator — JHU School Of Nursing
Locations (1):
- Johns Hopkins School of Nursing, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Ogungbe O, Hinneh T, Turkson-Ocran RN, Owusu L, Kumbe B, Spaulding EM, Gbaba S, Assani-Uva A, Mensah J, Yeboah-Kordieh Y, Sinyan A, Ampofo M, Oyedepo F, Commodore-Mensah Y. A Virtual Cardiometabolic Health Program Among African Immigrants in the US: A Pilot Cluster-Randomized Clinical Trial. JAMA Netw Open. 2025 Mar 3;8(3):e2462559. doi: 10.1001/jamanetworkopen.2024.62559. PMID 40036036